CLINICAL TRIAL: NCT03023046
Title: A Phase II Study of Dose-Adjusted Etoposide, Prednisone, Vincristine, Cyclophosphamide, and Doxorubicin (DA-EPOCH) as Front-Line Therapy for Adults With Acute Lymphoblastic Leukemia/Lymphoma
Brief Title: Etoposide, Prednisone, Vincristine Sulfate, Cyclophosphamide, and Doxorubicin in Treating Patients With Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ryan D. Cassaday, Associate Professor, Division of Hematology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9770; NCI-2016-02050 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9770 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1016012 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Results first posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Dasatinib; Doxorubicin; Etoposide; Imatinib Mesylate; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive etoposide IV over 96 hours, doxorubicin IV over 96 hours, and vincristine sulfate IV over 96 hours on days 1-4. Patients also receive cyclophosphamide IV over 1 hour on day 5 and prednisone PO BID on days 1-5. Patients who are Ph+ also receive imatinib mesylate or dasatinib PO QD on days 1-14. Patients who are CD20+ also receive rituximab IV on day 1 or day 5. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Dasatinib; Drug: Doxorubicin; Drug: Etoposide; Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; Cyclophosphamide Monohydrate
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel; 5-Thiazolecarboxamide; Dasatinib Hydrate; Dasatinib Monohydrate
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP57148B; Gleevec; Glivec; STI 571; STI-571; STI571
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83; Rituximab ABBS
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin (DA-EPOCH) works in treating patients with acute lymphoblastic leukemia or lymphoblastic lymphoma. Drugs used in chemotherapy, such as etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of either:

  * Acute lymphoblastic leukemia
  * Lymphoblastic lymphoma with detectable abnormal blasts in the bone marrow
* In the opinion of the treating investigator, patients must be an unsuitable candidate for a pediatric-inspired regimen, reasons for which may include (but not be limited to) older age (i.e., >= 40 years), practical/logistical barriers to or toxicity concerns from administration of a pediatric-inspired regimen, or Ph+ disease
* Total bilirubin =< 2.0 x institutional upper limit of normal ([ULN]; unless attributable to Gilbert's disease or other causes of inherited indirect hyperbilirubinemia, at which point total bilirubin must be =< 4.0 x ULN)
* Aspartate aminotransferases (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5.0 x institutional ULN; (Note: patients with liver test abnormalities attributable to hepatic involvement by ALL will be permitted if the total bilirubin is =< 5.0 x ULN and ALT/AST are =< 8.0 x ULN)
* Creatinine =< 2.0 mg/dL; however, patients with a creatinine > 2.0 mg/dL but with a calculated creatinine clearance of > 30 ml/min, as measured by the Modification of Diet in Renal Disease (MDRD) equation, will be eligible
* As patients with ALL frequently have cytopenias, no hematologic parameters will be required for enrollment or to receive the first cycle of treatment; however, adequate recovery of blood counts will be required to receive subsequent cycles)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2; (performance status of 3 will be allowed if poor performance status is thought to be directly secondary to ALL)
* Must agree to the use of effective contraception while on study treatment, unless they are highly unlikely to conceive (defined as [1] surgically sterilized, or [2] postmenopausal [i.e., a woman who is > 50 years old or who has not had menses for >= 1 year], or [3] not heterosexually active for the duration of the study)
* Ability to give informed consent and comply with the protocol
* Anticipated survival of at least 3 months, independent of ALL

Exclusion Criteria:

* Patients with Burkitt lymphoma/leukemia
* Patients must not have received any prior systemic therapy for ALL, except for the acute management of hyperleukocytosis or acute symptoms (e.g., corticosteroids, cytarabine, etc.)
* Patients with isolated extramedullary disease or with known parenchymal central nervous system (CNS) disease
* Known hypersensitivity or intolerance to any of the agents under investigation
* Other medical or psychiatric conditions that in the opinion of the investigator would preclude safe participation in the protocol
* May not be pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan D. Cassaday, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy)
Started | 54
Completed | 53
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 54 patients were consented and enrolled onto the study. 53 patients completed the study. 1 patient was not evaluable due to early treatment discontinuation.
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 53
Age, Continuous [Median (Full Range); unit: years] | 49 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
High white blood cell count [Count of Participants; unit: Participants] — A high white blood cell count is defined as greater than 30,000/uL for B-cell and greater than 100,000/uL for T-cell
  Participants | 11
Lineage [Count of Participants; unit: Participants]
  B-cell | 49
  T-cell | 4
Philadelphia chromosome [Count of Participants; unit: Participants] — Presence of Philadelphia chromosome, which is an abnormality of chromosome 22 in which part of chromosome 9 is transferred to it.
  Participants
    Philadelphia chromosome: positive | 28
    Philadelphia chromosome: negative | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Morphological Complete Response Rate
Description: Morphological complete remission (CR) was determined by bone marrow aspirate morphology and defined as <5% blasts by morphology, absolute neutrophil count >1000/uL, and platelet count >100,000/uL.
Time Frame: Within 4 cycles of study therapy
Measure: Count of Participants; unit: Participants
Groups:
- Ph+ Subjects: Subjects who have Philadelphia chromosome mutation
- Ph- Subjects: Subjects who do not have Philadelphia chromosome mutation
Arm/Group | Ph+ Subjects | Ph- Subjects
Number analyzed (Participants) | 28 | 25
Participants | 27 | 20

2. Primary Outcome: Number of Participants With Complete Measurable Residual Disease (MRD) Response Rate
Description: Response was determined by having no detectable disease by multiparameter flow cytometry (MFC-). For Ph+ subjects, complete molecular response (CMR) by BCR-ABL RT-PCR was assigned when MFC was undetectable.
  When no measurable residual disease was detected by MFC (MFC-) per EuroFlow criteria, high-throughput sequencing-based MRD testing (HTS; ClonoSEQ) was performed.
Time Frame: Within 4 cycles of study therapy
Population: HTS- percentages were calculated after excluding patients (Ph+, n = 4; Ph-, n = 3) that were unable to have HTS testing performed for technical reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph+ Subjects | Ph- Subjects
Number analyzed (Participants) | 28 | 25
Participants
  MFC-: Achieve within 4 cycles | 20 | 16
  MFC-: Not achieved within 4 cycles | 8 | 9
  CMR: number analyzed (Participants) | 28 | 0
  CMR: Achieve within 4 cycles | 11 |
  CMR: Not achieved within 4 cycles | 17 |
  HTS-: number analyzed (Participants) | 24 | 22
  HTS-: Achieve within 4 cycles | 8 | 6
  HTS-: Not achieved within 4 cycles | 16 | 16

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Grade 1 or higher non-hematologic adverse events will be assessed by Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Within 28 days of the last dose of the study drugs
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 53
Participants | 44

4. Secondary Outcome: Overall Survival
Description: Alive at 2 years after enrollment
Time Frame: Up to 2 years
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 53
Percentage of Participants | 70

5. Secondary Outcome: Event-free Survival
Description: Events were defined as any of the following: (1) unable to achieve either morphologic complete remission (CR) or MRD- by MFC, (2) relapse after CR, (3) MRD recurrence after achieving MRD-, or (4) death from any cause.
Time Frame: Up to 2 years
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment (Chemotherapy)
Number analyzed (Participants) | 53
Percentage of Participants | 32

ADVERSE EVENTS:
Time Frame: From the time patient signs consent through 30 days following discontinuation of study treatment, or until patient receives alternative anti-cancer therapy, whichever date comes first, up to 2 years.
Arm/Group | Treatment (Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 18/53
Serious Adverse Events (participants affected / at risk) | 32/53
Other Adverse Events (participants affected / at risk) | 14/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy) (N=53)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (19)
Fibrinogen decreased (Investigations) | 1 (1)
Fungemia (Infections and infestations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Kidney infection (Infections and infestations) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 9 (9)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy) (N=53)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The sample sizes in this study are relatively small, making it difficult to draw definitive conclusions regarding response rate and survival with this regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03023046/Prot_SAP_000.pdf